CLINICAL TRIAL: NCT04037826
Title: Randomized Clinical Trial on the Safety and Efficacy of L. Reuteri DSM 17938 and L. Reuteri ATCC PTA 6475 in the Treatment of Moderate to Severe Irritable Bowel Syndrome in Adults. Version 1.0, CSUB 0137, 27Jun2017
Brief Title: L. Reuteri DSM 17938 and L. Reuteri ATCC PTA 6475 in Moderate to Severe Irritable Bowel in Adults
Acronym: reuteri-IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovacion y Desarrollo de Estrategias en Salud (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Pedro Gutierrez Castrellon, Head of Research for Mother-Child, Innovacion y Desarrollo de Estrategias en Salud
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSUB 0137
Record Dates: First submitted 2019-07-27; First posted 2019-07-30 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome, adults, L. reuteri
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, controlled clinical trial, with two branches. Randomization will be centralized performed by sponsor. L. reuteri Gastrus at dose of 2x108 Colony Forming Units (CFU) or placebo will be adminsitrated twice per day
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be performed by Sponsor. Products will be send to research centers in blind bottles. Tablets for active and placebo have the same color and taste. Labelling will be performed in research centers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L. reuteri Gastrus (Experimental): L. reuteri Gastrus (L. reuteri DSM 17938 and L. reuteri ATCC PTA 6475)
  Interventions: Dietary Supplement: L. reuteri DSM 17938 and L. reuteri ATCC PTA 6475
- Placebo (Placebo Comparator): Placebo chewable tablets
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L. reuteri DSM 17938 and L. reuteri ATCC PTA 6475 — L. reuteri Gastrus (L. reuteri DSM 17938 and L. reuteri ATCC PTA 6475) at dose of 2x108 Colony Forming Units (CFU) per tablet. One chewable tablet is to be taken twice per day (one in the morning and one in the afternoon) giving a total daily dose of at least 4x108 CFU/day.
  Arms: L. reuteri Gastrus
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Randomized, double blind, controlled clinical trial, to evaluate safety and efficacy of L. reuteri DSM 17938 and L. reuteri ATCC PTA 6475 as adjuvant to reduce the severity of symptoms in adults with moderate to severe irritable bowel syndrome (IBS). Primary outcome: Global clinical Improve assessed by the GSRS-IBS score. Adults 18-65 years, any gender, with ROME IV criteria for moderate to severe IBS and body max index <36 will be included. Prescreening will be run for 2 weeks, the intervention period will be 2/days for 14t weeks, follow by a 2 weeks period of observation with no intervention. Secondary outcomes include: a) Improvements in the stool patterns evaluated through Bristol Stool Form (BSF); b) Improvement of the quality of life (QoL) measured by Latin-American IBS-QoL questionnaire; c) Improvement of the depression and anxiety severity evaluated by the Goldberg Depression and Anxiety Scale; d) Frequency of rescue medication use and e) Frequency of Adverse Events (AEs)

DETAILED DESCRIPTION:
Rationale: Irritable bowel syndrome (IBS) is the most commonly diagnosed functional gastrointestinal disorder observed in older children and adults. It is a frequent cause of chronic abdominal pain and changed bowel habits. Produce a significant negative effect on quality of life and it is associated with a significant economic burden disease con total expenditures in USA exceeding $20 billion/year. Since 2008 different clinical trials and meta-analysis had been published about the safety and efficacy of the use of probiotics in adults with IBS. In LATAM evidence about this topic is scarce.

Primary outcome: Global Clinical Improvement assessed by the GSRS-IBS score (Spanish/LA version) Secondary/Exploratory outcomes: Improvements in the Bristol Stool Form (BSF), Quality of Life (QoL) improvement assessed by Latin-American IBS-QoL questionnaire, Goldberg scale depression and Anxiety scale, Frequency of rescue medication use andSecondary adverse events Clinical design: Randomized, double blind, controlled clinical trial, with two arms Type of patients: Age 18-65 years, any gender, ROME IV diagnostic criteria for IBS (Recurrent abdominal pain, on average, at least 1 day per week in the last 3 months, associated with 2 or more of the following criteria a) Related to defecation, b) Associated with a change in frequency of stool, c) Associated with a change in form (appearance) of stool and/or d) Criteria fulfilled for the last 3 months with symptom onset at least 6 months before diagnosis), with a baseline GSRS-IBS score (Spanish/LA version) moderate to severe IBS, body mass index (BMI 25 to 35 (Mild to moderate obesity) and signed Informed consent.

Subject Information and Consent: All subjects will receive written and verbal information regarding the study at Visit 1. This information will emphasise that participation in the study is voluntary and that the subject may withdraw from the study at any time and for any reason. All subjects will be given the opportunity to ask questions about the study and will be given sufficient time to decide whether to participate in the study. Before any study-related procedures, the informed consent form will be signed and personally dated by the subject and by the person who conducted the informed consent discussion. A copy of the subject information including the signed consent form will be provided to the subject.

Interventions: 2 weeks run in, 14 weeks' treatment and 2 weeks follow up. L. reuteri Gastrus (L. reuteri DSM 17938 and L. reuteri ATCC PTA 6475) at dose of 2x108 Colony Forming Units (CFU). One chewable tablet is to be taken twice per day (one in the morning and one in the afternoon) giving a total daily dose of at least 4x108 CFU/day. The placebo will have identical ingredients except for lacking the bacteria. One chewable tablet is to be taken twice per day (one in the morning and one in the afternoon). The study products shall be kept refrigerated (+20C - +80C) during the study. Randomization will be performed by Sponsor Labelling will be performed in Research centres by independent pharmacist or similar person not involved in the study.

Study logistics: After informed consent, subjects must to fill a 2-week pre-randomization form to be sure they fill the criteria for IBS and define severity. If the patient fulfils all inclusion and none of the exclusion criteria the patient will be randomized to one of the two treatment groups. According to the randomization groups the patient will receive the corresponding blinded study product. The patient will be standardized to take the research product twice per day for 14 weeks, and complete the GSRS-IBS (Spanish/LA version) and the BSF on a daily basis, the Latin-American IBS-QoL questionnaire, the Goldberg depression and anxiety scale once, a diet history (2 days/week) and the report of adverse events. A basal faecal sample will be obtained in a subsample of patients to ultra-freeze and measure in a second-time microbiota by pyroseq and faecal calprotectin (At the end of treatment). At the end of treatment subjects will be evaluated according to primary and secondary/exploratory outcomes and they will be invited for a third periods, for 2 weeks with no intervention to evaluate the same clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Any gender
* ROME IV diagnostic criteria for IBS
* A baseline GSRS-IBS score (Spanish/LA version) moderate to severe IBS
* Body Mass Index (BMI) 25 to 35
* Patient capable of conforming to the protocol
* Signed Informed consent

Exclusion Criteria:

* Patients with relevant systemic, organic or metabolic diseases
* Patients with abnormal laboratory values that could be relevant to the outcome of study treatment
* Previous recent major abdominal surgery
* Consumption of antibiotics, Proton-Pump Inhibitors, H2-antagonists or dietary supplements containing Lactobacillus reuteri within 2 weeks prior to base-line
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Global clinical improvement | 16 weeks
  Global Clinical Improvement assessed by the GSRS-IBS score (Spanish/LA version). GSRS-IBS is a multidimensional score aimed to evaluate the severity of gastrointestinal IBS symptoms after and during treatment. It contains 13 items related to severity of abdominal pains, passing stools, abdominal tenderness, passing gas, constipation, diarrhea, etc. which had been validates in different languages.

SECONDARY OUTCOMES:
Improve on Stool Consistency | 16 weeks
  Improvements in the stool patterns evaluated through Bristol Stool Form (BSF). Bristol Scale is a validates score that evaluate the consistency of stools and classify the stools in 7 types (Type 1: separate hard lumps like nuts, type 2: sausage-shaped but lumpy and so on..)
Improve on Quality of Life | 16 weeks
  Improvement of the quality of life (QoL) measured by Latin-American IBS-QoL questionnaire. The IBS-QOL is a self-report quality-of-life measure specific to Irritable Bowel Syndrome (IBS) that can be used to assess the impact of IBS and its treatment. The IBS-QOL was developed using a needs based model. consists of 34 items, each with a five-point response scale. Items 1, 2, 4, 8-10, 12, 13, 16, 25-29, 34 are answered as 1. Not at all 2. Slightly 3. Moderately 4. Quite a bit 5. Extremely. Items 3, 5-7, 11, 14, 15, 17-24, 30-33 are answered as 1. Not at all 2. Slightly 3. Moderately 4. Quite a bit 5. A great deal. The different items are related how much the IBS impact QoL for subjects (i.e. 1. I feel helpless because of my bowel problems; 2. I am embarrassed by the smell caused by my bowel problems; 3. I am bothered by how much time I spend on the toilet, and so on...)
Improve on Depression | 16 weeks
  Improvement of the depression and anxiety severity evaluated by the Goldberg Depression and Anxiety Scale
Use of rescue medication | 16 weeks
  Frequency of use for rescue medication use
Adverse events | 16 weeks
  Frequency of Adverse Events after randomization (14 weeks during intervention and 2 weeks after stop intervention)

CONTACTS AND LOCATIONS:
Locations (2):
- Instituto de Nutricion y Tecnologia de los Alimentos, Santiago, Chile
- Hospital General Dr. Manuel Gea Gonzalez, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] McFarland LV, Dublin S. Meta-analysis of probiotics for the treatment of irritable bowel syndrome. World J Gastroenterol. 2008 May 7;14(17):2650-61. doi: 10.3748/wjg.14.2650. PMID 18461650
- [Result] Moayyedi P, Ford AC, Talley NJ, Cremonini F, Foxx-Orenstein AE, Brandt LJ, Quigley EM. The efficacy of probiotics in the treatment of irritable bowel syndrome: a systematic review. Gut. 2010 Mar;59(3):325-32. doi: 10.1136/gut.2008.167270. Epub 2008 Dec 17. PMID 19091823
- [Result] Tiequn B, Guanqun C, Shuo Z. Therapeutic effects of Lactobacillus in treating irritable bowel syndrome: a meta-analysis. Intern Med. 2015;54(3):243-9. doi: 10.2169/internalmedicine.54.2710. PMID 25748731
- [Result] Didari T, Mozaffari S, Nikfar S, Abdollahi M. Effectiveness of probiotics in irritable bowel syndrome: Updated systematic review with meta-analysis. World J Gastroenterol. 2015 Mar 14;21(10):3072-84. doi: 10.3748/wjg.v21.i10.3072. PMID 25780308
- [Result] Zhang Y, Li L, Guo C, Mu D, Feng B, Zuo X, Li Y. Effects of probiotic type, dose and treatment duration on irritable bowel syndrome diagnosed by Rome III criteria: a meta-analysis. BMC Gastroenterol. 2016 Jun 13;16(1):62. doi: 10.1186/s12876-016-0470-z. PMID 27296254